CLINICAL TRIAL: NCT03960359
Title: Inflammatory and Immune Profiles at the Time of a Severe Exacerbation in Preschool Asthmatic Children (<5 Years), According to the Phenotype
Brief Title: Inflammatory and Immune Profiles During a Severe Exacerbation in Preschool Asthmatic Children (<5 Years)
Acronym: VIRASTHMA2
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Région Nord-Pas de Calais, France (Other); Stallergenes Greer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014_20; 2014-A01687-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-17; First posted 2019-05-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Asthma; wheeze; preschool; phenotype
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, induced sputum, nasal swab sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic viral wheezers (EVW): EVW: Wheezing during discrete time periods (exacerbations), absence of symptoms between exacerbations Among which SIW: EVW with ≥ 2 exacerbations over the last 6 months Clinical, microbiological and inflammatory phenotype
  Interventions: Other: Clinical, microbiological and inflammatory phenotype
- Multiple trigger wheezers (MTW): MTW : wheezing during exacerbations but also symptoms between episodes. Clinical, microbiological and inflammatory phenotype
  Interventions: Other: Clinical, microbiological and inflammatory phenotype

INTERVENTIONS:
Other: Clinical, microbiological and inflammatory phenotype — Clinical phenotype: temporal pattern of wheeze (EVW, SIW, MTW), history and clinical data, allergy diagnosis work-up Microbiological phenotype: viral status (PCR in nasal swab sample), bacteriological status (culture of induced sputum) Inflammatory phenotype: profile of cytokines, phenotype of immune cells in the blood and the sputum, cytokine response to TLR ligands by peripheral blood mononuclear cells.

SUMMARY:
Asthma/wheeze begins in the first years of life and is the most common chronic disease in preschool children (< 5 years).

Different phenotypes have been suggested: Episodic-Viral Wheeze (EVW), absence of symptoms between exacerbations, among which Severe Intermittent Wheeze (SIW); and Multiple-trigger wheeze (MTW). The determinants of these different clinical phenotypes and their evolution have been poorly studied.

The purpose of this study is to assess preschool wheezers at the time of a severe exacerbation: clinical features and biological determinants (virus/bacteria, molecules and cells involved in the inflammation) and at steady state (8 weeks later) and to follow them up until the age of 7. The investigators hypothesize that the nature of the inflammation at the time of the exacerbation is different between these clinical phenotypes and may be associated with different clinical and functional trajectories

DETAILED DESCRIPTION:
Asthma/wheeze begins in the first years of life and is the most common chronic disease in preschool children (< 5 years).

Different phenotypes have been suggested: Episodic-Viral Wheeze (EVW): wheezing during discrete time periods (exacerbations), absence of symptoms between exacerbations; among which Severe Intermittent Wheeze (SIW): EVW with ≥ 2 exacerbations over the last 6 months; and Multiple-trigger wheeze (MTW): wheezing during exacerbations but also symptoms (cough, exercise-induced symptoms,…) between episodes. The determinants of these different clinical phenotypes and their evolution have been poorly studied.

The purpose of this study is to assess preschool asthmatic children at the time of a severe exacerbation: clinical features and biological determinants (virus/bacteria, molecules and cells involved in the inflammation) and at steady state (8 weeks later) and to follow them up until the age of 7. The investigators hypothesize that the nature of the inflammation at the time of the exacerbation is different between these clinical phenotypes and may be associated with different clinical and functional trajectories.

The primary objective is to compare levels of IFNg, IL-5, IL-13, IL-33, TSLP in blood and induced sputum between the 2 main phenotypes: EVW and MTW.

Preschool asthmatic children hospitalized for a severe exacerbation (requiring a course of systemic steroids) are included in a pediatric ward of one of the hospitals involved in the study, in the Hauts-de-France Region, France.

Clinical phenotype: temporal pattern of wheeze (EVW, SIW, MTW), history and clinical data, allergy diagnosis work-up Microbiological phenotype: viral status (PCR in nasal swab sample), bacteriological status (culture of induced sputum) Inflammatory phenotype: profile of cytokines, phenotype of immune cells in the blood and the sputum, cytokine response to TLR ligands by peripheral blood mononuclear cells will be assessed at the time of inclusion and at steady state 8 weeks later.

Children will be follow-up until the age of 7 (clinical data, control of asthma, lung function).

ELIGIBILITY:
Inclusion Criteria:

* Preschool children aged 1 to < 5 years
* Asthmatic / recurrent wheezers (≥ 3 discrete exacerbations since birth and/or symptoms between exacerbations, according to the definition from the French HAS and GINA guidelines)
* Hospitalized (less than 3 days ago) for a severe exacerbation (requiring a course of oral steroids)
* In a pediatric ward participating in the study (Hospital centers of Lille, Arras, Bethune, Douai, Lens, Roubaix, Tourcoing, Armentieres, Seclin)
* Parental consent

Exclusion Criteria:

* History of chronic disease (other than asthma)
* History of preterm birth (inf 36 weeks of amenorrhea)
* Lack of understanding from the parents

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preschool asthmatic children hospitalized for a severe exacerbation (requiring a course of systemic steroids), in a pediatric ward of one of the hospitals involved in the study, in the Hauts-de-France Region, France.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-02-24 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Inflammatory profile at exacerbation | At the time of the inclusion
  concentration levels of IFNg, IL-5, IL-13, IL-33, TSLP in blood and induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW

SECONDARY OUTCOMES:
Inflammatory profile at steady state | at baseline: consult at least 8 weeks after exacerbation
  concentration levels of IFNg, IL-5, IL-13, IL-33, TSLP in blood and induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Change of inflammatory profile between exacerbation and steady state | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  concentration levels of IFNg, IL-5, IL-13, IL-33, TSLP in blood and induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of cytokines in blood | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentration levels of cytokines (IL-4, IL-17A, IL-22, TNF-alpha, IL-1beta, IL-6, IL-10) in blood (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of cytokines in induced sputum | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentration levels of cytokines (IL-4, IL-17A, IL-22, TNF-alpha, IL-1beta, IL-6, IL-10) in induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of interferons in blood | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentrations levels of interferons (IFN-beta, IL-29) in blood (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of interferons in induced sputum | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentration levels of interferons (IFN-beta, IL-29) in induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of chemokines in blood | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentration levels of chemokines (CXCL8, CXCL10, CCL5, CCL20) in blood (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Levels of chemokines in induced sputum | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Concentration levels of chemokines (CXCL8, CXCL10, CCL5, CCL20) in induced sputum (all concentrations expressed in pg/ml, obtained with multiplex assays) between wheeze patterns: EVW (among which SIW) vs MTW
Expression patterns of mononuclear cells | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Percentage of mononuclear cells in peripheral blood and sputum (sorted by flow cytometry): lymphocytes, dendritic cells, innate lymphoid cells
Percentage of patients with tobacco exposure | At the time of the inclusion
  Percentage of tobacco exposure (qualitative data)
Percentage of patients with mould/moisture exposure | At the time of the inclusion
  Percentage of visible mould/moisture exposure (qualitative data, based on declaration by the parents)
Percentage of patients with pet ownership | At the time of the inclusion
  Percentage of pet ownership (qualitative data)
Percentage of patients living in urban area | At the time of the inclusion
  Percentage of urban living (qualitative data)
number of asthma exacerbations in the previous year | At the time of the inclusion
  number of asthma exacerbations in the previous year (quantitative data)
Percentage of patients with associated atopic diseases | At the time of the inclusion
  Percentage of associated atopic disorders: atopic dermatitis, atopic rhinitis, food allergy (qualitative data)
Control of asthma | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Control of asthma based on symptoms (breath, cough, breathlessness, impact on activity and social behavior) and previous exacerbations in the past year, and classified according to GINA criteria: well-controlled, partly controlled, uncontrolled (semi-quantitative)
Features of the exacerbation: severity | At the time of the inclusion
  Severity assessed during the first hour in the emergency department (before treatment), using PRAM severity score: mild asthma (0-3), moderate asthma (4-7), severe asthma (8-12) (quantitative data)
Features of the exacerbation: length | At the time of the inclusion
  Length of stay and length of oxygen need (in days)
Atopy | At the time of the inclusion and at the age of 7
  Atopy: positivity of skin prick tests (≥ 3 mm diameter) and/or specific IgE (≥ 0,35 ku/l), mono or polysensitized status (qualitative data)
Blood leukocyte count | At the time of the inclusion and at the age of 7
  Count of neutrophils and eosinophils (number/mm3)
ImmunoCAP ISAC (Thermo Fisher Scientific) | At the time of the inclusion and at the age of 7
  Levels of component specific IgE antibodies will be expressed in ISAC standardized units (ISU). We will categorized the raw data into 4 sIgE semiquantitative discrete groups, according to the manufacturer's guidelines: no (<0.3 ISU), low (0.3-1 ISU), medium (1-15 ISU), and high (>15 ISU) sensitization
Microbiological phenotype: viral status | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Virus identification by PCR in nasal swab sample (qualitative data)
Microbiological phenotype: bacteriological status | At the time of the inclusion and at baseline (consult at least 8 weeks after exacerbation)
  Positive identification of bacteria (positive if titer >= 10.4/ml) by culture of induced sputum (qualitative data)
History at the age of 7 | At the age of 7
  History of asthma exacerbations in the previous year, presence of other atopic diseases: atopic dermatitis, atopic rhinitis, food allergy (qualitative data)
Control of asthma at the age of 7 | At the age of 7
  Control of asthma based on symptoms (breath, cough, breathlessness, impact on activity and social behavior) and previous exacerbations in the past year, and classified according to GINA criteria: well-controlled, partly controlled, uncontrolled (semi-quantitative)
Atopy at the age of 7 | At the age of 7
  Atopy: positivity of skin prick tests (≥ 3 mm diameter) and/or specific IgE (≥ 0,35 ku/l), mono or polysensitized status (qualitative data)
Lung function at the age of 7: forced expiratory volume in one second | At the age of 7
  Forced expiratory volume in one second (FEV1) after administration of short acting beta agonists, obtain with spirometry test (expressed in Z-score)
Lung function at the age of 7 : forced vital capacity | At the age of 7
  Forced vital capacity (FVC) after administration of short acting beta agonists, obtain with spirometry test (expressed in Z-score)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Deschildre, MD, Principal Investigator — University Hospital, Lille